CLINICAL TRIAL: NCT02602444
Title: Comparison of Ticagrelor Pharmacokinetics and Pharmacodynamics in ST-elevation Myocardial Infarction and Non-ST-elevation Myocardial Infarction Patients
Brief Title: Comparison of Ticagrelor Pharmacokinetics and Pharmacodynamics in STEMI and NSTEMI Patients
Acronym: PINPOINT
Status: Completed | Type: Observational
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. dr hab., Collegium Medicum w Bydgoszczy
Other Study IDs: CMUMK202B
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Myocardial Infarction
Keywords: ticagrelor; STEMI; NSTEMI; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STEMI: ST-elevation myocardial infarction patients receiving 180 mg ticagrelor loading dose
  Interventions: Drug: ticagrelor
- NSTEMI: non-ST-elevation myocardial infarction patients receiving 180 mg ticagrelor loading dose
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — 180 mg loading dose
  Other Names: Brilique

SUMMARY:
The purpose of the PINPOINT study is to compare pharmacokinetics (PK) and pharmacodynamics (PD) of ticagrelor in ST-elevation myocardial infarction (STEMI) and non-ST-elevation myocardial infarction (NSTEMI) patients designated to invasive strategy. Data regarding comparison of PK and antiplatelet action of ticagrelor in STEMI and NSTEMI are sparse. Recommended dosing regimens of ticagrelor are identical for both STEMI and NSTEMI, although it is not known whether PK and PD features of ticagrelor are uniform in these patients.

DETAILED DESCRIPTION:
The European Society of Cardiology and American Heart Association guidelines recommend use of ticagrelor or prasugrel as a treatment of choice in patients with both STEMI and NSTEMI (class of recommendation I, level of evidence B). Recommended dosing regimens of ticagrelor are identical in STEMI and NSTEMI patients, although epidemiology, clinical approach and early outcomes differ between these two types of myocardial infarction. It is not known whether PK and PD features of ticagrelor are uniform in STEMI and NSTEMI patients. However, the existing body of evidence suggest that PK and PD of ticagrelor may be attenuated in STEMI patients compared to healthy subjects and patients with stable coronary artery disease, which may expose STEMI patients at increased risk of developing thrombotic complications secondary to insufficient platelet inhibition. The PINPOINT study could provide a valuable insight into the knowledge regarding ticagrelor action in STEMI vs. NSTEMI patients.

Since there is no reference study comparing pharmacokinetics of ticagrelor in STEMI and NSTEMI patients, we decided to perform an internal pilot study of approximately 30 patients (15 patients with each type of myocardial infarction) for estimating the final sample size.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent prior to any study specific procedures
* diagnosis of acute ST-segment elevation myocardial infarction or acute non-ST-segment elevation myocardial infarction
* male or non-pregnant female, 18 years old and older
* provision of informed consent for angiography and PCI

Exclusion Criteria:

* treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* hypersensitivity to ticagrelor
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* active bleeding
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of coagulation disorders
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* second or third degree atrioventricular block during screening for eligibility
* patient required dialysis
* manifest infection or inflammatory state
* Killip class III or IV during screening for eligibility
* respiratory failure
* current therapy with strong CYP3A inhibitors or strong CYP3A inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI or NSTEMI admitted to the study centre, designated to invasive strategy.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve for ticagrelor (AUC 0-6h) | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h post dose

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve for AR-C124910XX (AUC 0-6h) | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h post dose
Area under the plasma concentration-time curve for ticagrelor (AUC 0-12h) | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h, 12h post dose
Area under the plasma concentration-time curve for AR-C124910XX (AUC 0-12h) | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h, 12h post dose
Maximum concentration (Cmax) of ticagrelor and AR-C124910XX | 12 hours
Time to maximum concentration (Cmax) for ticagrelor and AR-C124910XX | 12 hours
Platelet reactivity index (PRI) assessed by VASP assay | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h, 12h post dose
Platelet reactivity assessed by Multiple Electrode Aggregometry | prior to the initial dose and 30min, 1h, 2h, 3h, 4h, 6h, 12h post dose
  It will be assessed in all predefined time points in all study participants except those treated with GP IIb/IIIa receptor inhibitors.
Percentage of patients with high platelet reactivity (HPR) after the loading dose of ticagrelor assessed with VASP and Multiple Electrode Aggregometry | 2 hours
Time to reach platelet reactivity below the cut-off value for HPR evaluated with VASP and Multiple Electrode Aggregometry | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

REFERENCES:
- [Derived] Adamski P, Sikora J, Laskowska E, Buszko K, Ostrowska M, Uminska JM, Sikora A, Skibinska N, Sobczak P, Adamska U, Rosc D, Kubica A, Paciorek P, Marszall MP, Navarese EP, Gorog DA, Kubica J. Comparison of bioavailability and antiplatelet action of ticagrelor in patients with ST-elevation myocardial infarction and non-ST-elevation myocardial infarction: A prospective, observational, single-centre study. PLoS One. 2017 Oct 12;12(10):e0186013. doi: 10.1371/journal.pone.0186013. eCollection 2017. PMID 29023473
- [Derived] Adamski P, Ostrowska M, Sikora J, Obonska K, Buszko K, Krintus M, Sypniewska G, Marszall MP, Kozinski M, Kubica J. Comparison of Ticagrelor Pharmacokinetics and Pharmacodynamics in STEMI and NSTEMI Patients (PINPOINT): protocol for a prospective, observational, single-centre study. BMJ Open. 2017 Apr 26;7(4):e013218. doi: 10.1136/bmjopen-2016-013218. PMID 28446521